CLINICAL TRIAL: NCT05348967
Title: Association of D-chiro-inositol and the Ketogenic Diet in the Treatment of Overweight/Obese Patients With Insulin Resistance and Polycystic Ovary Syndrome
Brief Title: Combination of D-chiro-inositol With Ketogenic Diet
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No partecipants enrolled
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCI_KETO22
Record Dates: First submitted 2022-04-22; First posted 2022-04-27 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Ketogenic diet
- TECADRIOL (Experimental): Ketogenic diet plus a food supplement containing an association of D-chiro-inositol and alpha-lactalbumin
  Interventions: Dietary Supplement: TECADRIOL

INTERVENTIONS:
Dietary Supplement: TECADRIOL — Food supplement with D-chiro-inositol and alpha-lactalbumin
  Arms: TECADRIOL

SUMMARY:
The study aims to evaluate whether the combination of a product based on D-chiro-inositol and the ketogenic diet can improve the metabolic/endocrine picture of overweight/obese women with PCOS, with insulin resistance, in a shorter time than the ketogenic diet alone

DETAILED DESCRIPTION:
Weight loss is the main approach to counteract PCOS phenotype, improving ovulatory function and reducing insulin and systemic levels of free testosterone.

It is not yet ascertained whether the composition of the diet can have a positive effect on the metabolic pattern; however, it should be considered that blood glucose levels are influenced by the intake of carbohydrates that regulate insulin secretion.

Therefore, low-carbohydrate diets should be preferred over standard low-calorie diets, in terms of improvement in metabolic/endocrine parameters, which accompanies weight loss in women with PCOS.

The ketogenic diet (KD), a very low-carbohydrate diet capable of developing physiological ketosis, has proven very effective aganist various pathological conditions, including obesity and type 2 diabetes.

In particular, in the context of KD there is an ever increasing interest in VLCKD (Very Low Calorie Ketogenic Diet) diets with very low calorie content as well as carbohydrates, which have been shown to be effective and safe in the management of metabolic diseases.

Evidence on the efficacy of this diet in PCOS women is still rather scarce. An uncontrolled pilot study, in which VLCKD was followed by 11 overweight/obese women with PCOS for a period of 24 weeks, demonstrated a significant reduction in body weight, free testosterone, LH to FSH ratio and, especially, fasting insulin, suggesting favorable effects in PCOS patients.

It has been widely demonstrated that the supplementation of inositols, polyols with insulin-sensitizing action, can normalize the metabolic/endocrine picture of PCOS patients, who are overweight/obese and insulin resistant, avoiding the typical gastrointestinal side effects of classic insulin sensitizers.

A recent study on overweight/obese women with PCOS has shown that the association of (low-calorie) diet with inositol supplementation accelerates weight loss, contributing to the restoration of the menstrual cycle.

Therefore, considering the results of this study and bearing in mind the literature that reports that D-chiro-inositol improves glucose tolerance and increases insulin sensitivity in hyperinsulinemic women with polycystic ovary syndrome, we want to investigate whether supplementation with D-chiro-inositol in association with VLCKD can improve the metabolic/endocrine profile of overweight/obese insulin resistant PCOS women in a shorter time than with VLCKD alone.

This would reduce the period in which patients undergo the VLCKD diet, allowing them to follow a less restrictive and subsequently maintenance diet in the shortest possible time.

ELIGIBILITY:
Inclusion Criteria:

* Women with age between 25 and 40 years
* Diagnosis of Polycystic Ovary Syndrome (PCOS)
* Diagnosis of insulin-resistance (HOMA ≥2.5)
* 26 ≤ BMI ≤32

Exclusion Criteria:

* Subjects with no indication for treatment
* Pregnancy, breastfeeding
* Treatment with drugs or supplements that interfere with the mechanism of action of insulin

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
HOMA index | Three time points: change in HOMA index from the baseline to 2 and 4 months
  Reduction of HOMA index

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No